CLINICAL TRIAL: NCT06516913
Title: A Randomized, Participant-Blinded Study to Investigate the Effects of Subcutaneous Injection Volume, Injection Rate, and Needle Length on Pain in Healthy Participants
Brief Title: A Study of Subcutaneous Injection in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 27209; J3G-MC-S004 (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (8):
- Sequence 1 (ABHCGDFE) (Experimental): Syringe pump is used to subcutaneously (SC) administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 2 (BCADHEGF) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 3 (CDBEAFHG) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 4 (DECFBGAH) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 5 (EFDGCHBA) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 6 (FGEHDACB) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 7 (GHFAEBDC) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump
- Sequence 8 (HAGBFCED) (Experimental): Syringe pump is used to SC administer buffer solution with hyaluronic acid as a viscosity agent
  Interventions: Device: Harvard Apparatus syringe pump

INTERVENTIONS:
Device: Harvard Apparatus syringe pump — Used to administer buffer solution with hyaluronic acid SC.

SUMMARY:
This is a device feasibility study designed to evaluate the practicality of delivering a high-viscosity solution subcutaneously using various injection parameters, including volume, rate, and needle length. The goal is to assess the usability and operational performance of a delivery setup (Havard apparatus syringe pump and related components) to inform design requirements for future large-volume injection devices.

No active drug is administered in this study, and no health outcomes are being evaluated.

The study duration is approximately 40 days, including screening, injection assessments, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy as determined by medical evaluation including medical history and physical examination
* Have a waist circumference, measured around umbilicus, of at least 78 centimeters (cm) for participants assigned male at birth, and at least 71 cm for participants assigned female at birth
* Have a BMI within the range of 21.0 to 30.0 kilograms per square meter (kg/m²)
* Participants assigned female at birth must be of non-childbearing potential and must test negative for pregnancy prior to injection on Day 1

Exclusion Criteria:

* Have known allergies to hyaluronic acid, related compounds, or any components of the formulation, or history of significant atopy. Components of the formulation include, but are not limited to, sodium hyaluronate, sodium chloride, and sodium phosphate
* Have a history of severe injection-site reactions
* Have current or previous history of anaphylaxis
* Have tattoos or scars over the abdomen, or other factors, for example excessive folds of skin, that, in the investigator's opinion, would interfere with injection site assessments
* Have self-perceived dullness or loss of sensation on either side of the body and the abdomen
* Have a history or presence of a bleeding, wound healing (including diabetes), or fibrotic disorder
* Have known or ongoing psychiatric disorders

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Usability Assessment of Subcutaneous Injections Using a Syringe Pump Across Multiple Delivery Parameters | Day 1
  Usability will be assessed by evaluating the proportion of subcutaneous injections administered using Harvard Apparatus syringe pump across varying injection volumes, rates, and needle lengths.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea CRU, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No